CLINICAL TRIAL: NCT01616264
Title: Evaluation of the Reproducibility of Computed Tomography for the Measurement of Tuberculosis Pleural Effusion
Brief Title: Reproducibility of Computed Tomography
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Juliana Flávia de Oliveira, Phd, Universidade Federal do Rio de Janeiro
Other Study IDs: JUL 200456
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Tuberculosis; Pleural Effusion
Keywords: Tuberculosis; Pleural Effusion; Computed Tomography
MeSH Terms: conditions — Tuberculosis; Pleural Effusion

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Thus, the aim of this study was to evaluate the reproducibility of the Computed Tomograph scan three-dimensional reconstruction method for the measurement of the TB pleural effusion volume in clinically stable patients.

DETAILED DESCRIPTION:
Speed, accuracy, and precision in the quantification of pleural effusion are of critical importance as it determines whether or not thoracocentesis should be carried out and which technique should be employed for such a procedure. This study evaluates the precision of thoracic computed tomography with three-dimensional (3D) rebuilding in determining the volume of tuberculosis pleural effusion.Twenty patients with pleural effusion were screened and invited to take part in the study. Each patient underwent two computed tomography scans, before and after one month of treatment for tuberculosis, a total of 40 exams. These were evaluated by two expert radiologists. In conclusion, the quantification of the pleural effusion volume by using thoracic CT with volumetric three-dimensional reconstruction is a highly reproducible method.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years with a confirmed diagnosis of pleural TB effusion .
* Signed out an informed consent term

Exclusion Criteria:

* Patients with human immunodeficiency virus (HIV).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 years or older with a confirmed diagnosis of pleural TB effusion
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana F Oliveira, Phd, Principal Investigator — Universidade Federal do Rio de Janeiro